CLINICAL TRIAL: NCT00034801
Title: A Controlled Trial of Olanzapine Versus Active Comparator in the Treatment of Schizophrenic and Schizoaffective Subjects With Comorbid Depression
Brief Title: Olanzapine Versus Active Comparator in the Treatment of Depression in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5529; F1D-US-HGJU
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Depression; Schizophrenia; Schizoaffective Disorder
Keywords: Depression; Comorbid Depression; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Depression; Schizophrenia; Psychotic Disorders | interventions — Olanzapine; ziprasidone

INTERVENTIONS:
Drug: olanzapine
Drug: ziprasidone

SUMMARY:
This is a research study comparing the safety and efficacy of two active study medications

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-60 years of age
* Female subjects of childbearing potential must be using a medically accepted means of contraception
* Each subject must have a level of understanding sufficient to perform all tests and examinations required by the protocol
* Subjects must be considered reliable

Exclusion Criteria:

* Treatment with a drug within the last 30 days that has not received regulatory approval at the time of study entry
* Female subjects who are either pregnant or nursing
* Uncorrected hypothyroidism or hyperthyroidism
* Narrow-angle glaucoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 378
Dates: Start 2001-09; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Tuscaloosa, Alabama
  - Little Rock, Arkansas
  - Anaheim, California
  - Chula Vista, California
  - Lafayette, California
  - Long Beach, California
  - Orange, California
  - Poway, California
  - Rosemeade, California
  - San Diego, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Winter Park, Florida
  - Augusta, Georgia
  - Prairie Village, Kansas
  - Gaithersburg, Maryland
  - Mount Pleasant, Michigan
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Clementon, New Jersey
  - Buffalo, New York
  - New York, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Sioux Falls, South Dakota
  - Austin, Texas
  - El Paso, Texas
  - Houston, Texas
  - Salt Lake City, Utah